CLINICAL TRIAL: NCT05386121
Title: Ultrasound Guided Erector Spinae Plane Block Versus Quadratus Lumborum Block in Pediatric Open Renal Surgeries: A Randomized Comparative Study.
Brief Title: Erector Spinae Plane Block Versus Quadratus Lumborum Block for Open Renal Surgeries in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kareem Mohammed Assem Nawwar, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: md-13-2022
Record Dates: First submitted 2022-05-08; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl; Meperidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector spinae plane block (ESPB) group (Active Comparator): 30 child will receive a preoperative unilateral single shot US-guided erector spinae plane block at the level of T9 vertebra in the lateral position after induction of general anesthesia, using 0.5 mL/kg of bupivacaine 0.125%
  Interventions: Procedure: Ultrasound-guided Erector Spinae Plane Block; Device: Ultrasound Machine; Device: Echogenic needle; Drug: Fentanyl; Drug: Pethidine
- Quadratus lumborum block (QLB) group (Active Comparator): 30 child will receive a preoperative unilateral single shot US-guided quadratus lumborum block at the level of L2 spinous process in the lateral position after induction of general anesthesia, using 0.5 mL/kg of bupivacaine 0.125%
  Interventions: Procedure: Ultrasound-guided Quadratus Lumborum Block; Device: Ultrasound Machine; Device: Echogenic needle; Drug: Fentanyl; Drug: Pethidine

INTERVENTIONS:
Procedure: Ultrasound-guided Erector Spinae Plane Block — Using a 22-gauge 80 mm echogenic needle under ultrasound guidance, 0.5 mL/kg of bupivacaine 0.125% will be injected in the fascial plane deep to erector spinae muscle after conﬁrming correct needle location by a negative aspiration test then by injecting 0.5-1 ml saline and observing the ﬂuid lifting the erector spinae muscle off the transverse process (hydrodissection). The ultrasound probe will be placed 2-3 cm lateral to the spinous process on a parasagittal plane, to visualize the erector spinae muscle and transverse process, directing the needle craniocaudally using the in-plane technique. The spread of the injectate will be observed to distribute within this plane.
  Arms: Erector spinae plane block (ESPB) group
Procedure: Ultrasound-guided Quadratus Lumborum Block — Using a 22-gauge 80 mm echogenic needle under ultrasound guidance, 0.5 mL/kg of bupivacaine 0.125% will be injected in the fascial plane between the quadratus lumborum and psoas major muscle after conﬁrming correct needle location by a negative aspiration test then by injecting 0.5-1 ml saline (hydrodissection). The ultrasound probe will be placed 2-3 cm lateral to the L2 spinous process on an axial plane, to visualize the transverse process with psoas major muscle anterior, quadratus lumborum muscle lateral and erector spinae muscle posterior to it. The needle is inserted from the medial side of the probe and advanced laterally using the in-plane technique. The spread of the injectate will be observed to distribute within the target plane.
  Arms: Quadratus lumborum block (QLB) group
Device: Ultrasound Machine — Sonosite S-Nerve (USA) with a linear multi-frequency 6-13 MHz (hockey stick) transducer
Device: Echogenic needle — A 22-gauge 80 mm needle the sonoplex needle manufactured by PAJUNK (USA)
Drug: Fentanyl — Given intravenously (1 µg/kg) as part of induction of general anesthesia (GA) added to propofol 2 mg/kg and atracurium 0.5 mg/kg Intraoperatively, intravenous fentanyl 0.5 µg/kg (with a maximum dose of 2 µg/kg) will be administered in response to any increase in hemodynamics by more than 20% of baseline values in response to skin incision or there after throughout surgery (after exclusion of other causes of hemodynamic changes)
Drug: Pethidine — Will be given intravenously as a rescue analgesic (0.5 mg/kg with maximal dose 1.5 mg/kg) in both study groups if Children's Hospital Eastern Ontario Pain Scale (CHEOPS) more than 6. Quality of postoperative analgesia will be assessed using CHEOPS pain score at time transfer to PACU, 15, 30 minutes then 1, 2, 4, 6 hours postoperatively.

SUMMARY:
Open renal surgeries are associated with significant postoperative pain; early control of the perioperative pain is associated with decrease of hemodynamic variations during the surgery, early mobilization, better quality of functional recovery & early discharge of patients. Side effects of systemic opioids, as well as difficulty to monitor their response, are major limitations to their use.

Pediatric regional anesthesia (PRA) is one of the most valuable and safe tools to treat perioperative pain, and is an essential part of modern anesthetic practice. Neuraxial analgesia for pediatric patients is a mode of pain control that gained popularity in the last few decades as it decreases opioid exposure, shortens recovery room time & hospital stay. Caudal block is the most commonly used neuraxial anesthesia in pediatric patients. However, its major side effect is urinary retention and excessive motor block.

Considerable progress has been made in the practice of PRA over the past few years including incorporation of ultrasound guidance, with promising novel regional anesthesia techniques, especially the anterolateral and the posterolateral trunk blocks.

In this study, the investigators will compare the ultrasound guided quadratus lumborum block (QLB) with erector spinae plane block (ESPB), regarding the duration and quality of postoperative analgesia in pediatric patients undergoing unilateral open renal surgeries under general anesthesia. The study hypothesis is that QLB can provide a more superior postoperative pain relief to ESPB in children undergoing open renal surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. American society of anesthesiologists (ASA) class I and II
2. Children undergoing unilateral open renal surgeries

Exclusion Criteria:

1. Parents refusal for the block
2. Bleeding disorders (platelets count < 100,000/uL; INR > 1.5; PC < 60%)
3. Skin lesion, wounds or infection at the puncture site.
4. Known allergy to local anesthetic drugs

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Time to first postoperative rescue analgesia | 12 hours
  Time in minutes when postoperative Children's Hospital Eastern Ontario Pain Scale (CHEOPS) pain score exceeds 6 for the first time. Children's Hospital Eastern Ontario Pain Scale is a pain score with the least possible score is 4, while the highest possible score 13 (worse outcome).

SECONDARY OUTCOMES:
Total opioid analgesic consumption in the first 12 hours postoperative period | from time of patient transfer to the PACU, till 12 hours postoperatively
  when postoperative Children's Hospital Eastern Ontario Pain Scale (CHEOPS) pain score ˃ 6 in the first 12 hours postoperatively. Children's Hospital Eastern Ontario Pain Scale is a pain score with the least possible score is 4, while the highest possible score 13 (worse outcome).
Intraoperative mean arterial blood pressure | During surgery (from induction of general anesthesia till 15 mins. after performance of the nerve block)
  measured from induction of general anesthesia, after performance of the nerve block and at 1,5,10, 15 mins. after
Intraoperative heart rate | During surgery (from induction of general anesthesia till 15 mins. after performance of the nerve block)
  measured before and after induction of general anesthesia, after performance of the nerve block and at 1,5,10, 15 mins. after
Postoperative pain score | from time of patient transfer to the PACU, till 12 hours postoperatively
  measured at time of patient transfer to the PACU, 15, 30 mins, 1 ,2 , 4 ,6 ,12 hours after surgery
Block performance time | Time from ultrasound visualization of target injection site to end of local anesthetic (bupivacaine) deposition up to 15 mins.
  Time to perform ultrasound guided nerve block

OTHER OUTCOMES:
Indirect signs of local anesthetic toxicity | from time of local anesthetic (bupivacaine) deposition till 6 hours postoperatively
  intraoperative arrhythmias and delayed awakening

CONTACTS AND LOCATIONS:
Overall Officials: Nevine M Gouda, Study Chair — Cairo University; Sherif M Soaida, Study Chair — Cairo University; Ismail S Hammad, Study Chair — Cairo University; Ahmed T Bahnaswy, Principal Investigator — Cairo University